CLINICAL TRIAL: NCT03716908
Title: Evaluation of Hearing and Vestibular Function in Presymptomatic and Symptomatic DFNA9 Patients Carrying the Pro51Ser (P51S) Mutation in the COCH Gene.
Brief Title: Genotype-phenotype Correlation Study of Presymptomatic and Symptomatic DFNA9 Patients
Status: Recruiting | Type: Observational
Sponsor: Jessa Hospital (Other)
Collaborators: University Hospital, Antwerp (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: JessaHORL2
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-08

CONDITIONS: Vestibular Diseases; DFNA9
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood samples for the genetic diagnosis of carriership of P51S COCH mutation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P51S+ group: Group 1 affected subjects (P51S+) Family member P51S mutation carrier
  interventions/ Questionnaire (DHI, OS, EQ-D5-5L, ABC) Pure Tone audiometry VNG vHIT c- and o-VEMP
- P51S- group (healthy control): Group 2: healthy control Family member P51S non-carrier
  interventions: Questionnaire (DHI, OS, EQ-D5-5L, ABC) Pure Tone audiometry VNG vHIT c- and o-VEMP

SUMMARY:
DFNA9 (Deafness Autosomal Dominant 9) is an autosomal dominant hereditary hearing loss which is associated with vestibular deterioration. The most recent genotype-phenotype correlation studies have been conducted more than 15 years ago. Meanwhile, emerging and valuable vestibular tests have been added to the vestibular test battery. These tests were not available at the time of the correlation studies. The aim of this study is to carry out a prospective cross-sectional study on symptomatic and presymptomatic affected carriers of the Pro51Ser (P51S) Coagulation Factor C Homology (COCH) mutation in order to correlate vestibular data using the complete vestibular test battery with the known data on hearing and vestibular function in relation to age.

DETAILED DESCRIPTION:
Systematic review of the genotype-phenotype correlation studies in P51S carriers has shown an underrepresentation of presymptomatic affected subjects and the calculation of vestibular deterioration were based on just one vestibular parameter, whereas the combined evaluation of a complete vestibular test battery, covering the complete vestibular sensitivity range and all labyrinthine compartments separately, is nowadays considered standard practice in determining more accurate assessment of the vestibular function.

For this reason, a prospective cross-sectional study on pre- as well as symptomatic DFNA9 patients carrying the Pro51Ser (P51S) mutation in COCH gene is being carried out, in order to gain more realistic data on vestibular dysfunction, consisting of pure tone audiometry and a comprehensive vestibular test battery, including electro- or videonystagmography (VNG), C- and O-Vestibular-evoked myogenic potential (VEMP) tests, video Head Impulse Test (vHIT) and questionnaires (DHI (Dizziness handicap Index), oscillopsia questionnaire (OS), Quality of Life Questionnaire (EQ-5D-5L), activities-specific balance confidence (ABC) scale.

ELIGIBILITY:
Inclusion Criteria:

* subject must be 18 year of older
* subject is a family member of the family pedigree's proband(s) carrying a P51S COCH mutation

Exclusion Criteria:

* subject is younger than 18 years
* subject is not a family member of the pedigree's proband(s) carrying a P51S
* subject cannot undergo investigations (medical and/or mental reasons)
* subject is not willing to be enrolled into the study
* subject suffers other concomitant middle or inner ear disease
* subject has undergone middle ear or inner ear surgery
* subject suffers other concomitant vestibular disease than DFNA9
* subject has undergone vestibular surgery or other non-invasive vestibular treatment (gentamicin intratympanal injections for example)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all family pedigree in which at least one proband is carrying the Pr51Ser (P51S) mutation in the COCH gene that are known in three tertiary referral centers: University Hospital Antwerp, Maastricht University Medical Centre and Jessa Hospital Hasselt.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
hearing threshold | 1 year
  pure tone audiometry, decibel hearing loss (dB HL)
video HIT | 1 year
  video Head Impulse test, gain (eye movement versus head movement)

SECONDARY OUTCOMES:
VEMP | 1 year
  c- and o-VEMP tests (vestibular-evoked myogenic potentials): threshold (decibel sound pressure level: dB SPL or dB HL)
DHI questionnaire | 1 year
  DHI (dizziness handicap index): scores the degree of imbalance perception of the patient, the higher the score, the higher the imbalance perception; normative score below 10
OS questionnaire | 1 year
  A questionnaire assessing oscillopsia severity for patients with bilateral vestibulopathy and patients with unilateral vestibular lesions. Oscillopsia was defined as a "sensation that the visual environment is moving when it's not." The 9-item questionnaire investigates oscillopsia frequency in different situations encountered in daily life. Each item was scored 1 (never), 2 (seldom), 3 (sometimes), 4 (often), or 5 (always). Scores were averaged to provide an oscillopsia severity score ranging from 1 to 5. A mean score higher than 3 is considered to indicate moderate to extreme oscillopsia severity.
ABC questionnaire | 1 year
  ABC activities specific balance confidence scale to asses individual's confidence in performing daily activities , scores from 0-100%, normative values >80%
EQ-5D-5L questionnaire | 1 year
  Quality of life questionnaire:EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal; 5 dimensions: anxiety/depression, discomfort/pain, usual activities, mobility and self-care are evaluated in 5 levels (ranging from no problems (level 1) to extreme problems (level 5) and a Vertical Visual Analogue Scale (VAS) EQ-VAS ranging from 0 (worst health) to 100 (best health), convertible to an index value. result presentation in EQ-5D (dimensions), EQ-VAS and EQ-5D-5L index values with normative values per age group, all as a measure of central tendency and a measure of dispersion using mean values and standard deviation per age group
Caloric response | 1 year
  Caloric response using 4 successive water irrigation at 30 and 44 degrees Celsius , summation of the gain of the slow phase of the elicited nystagmus of all 4 irrigations (degrees per second) , normative values to be established for each vestibular laboratory in healthy control subjects
SHAT | 1 year
  Sinusoidal harmonic acceleration test (SHAT) of rotatory chair in the dark with open eyes, degrees per second, normative values to be established for each vestibular laboratory on healthy control subjects

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] JanssensdeVarebeke SPF, Moyaert J, Fransen E, Bulen B, Neesen C, Devroye K, van de Berg R, Pennings RJE, Topsakal V, Vanderveken O, Van Camp G, Van Rompaey V. Genotype-Phenotype Correlation Study in a Large Series of Patients Carrying the p.Pro51Ser (p.P51S) Variant in COCH (DFNA9) Part II: A Prospective Cross-Sectional Study of the Vestibular Phenotype in 111 Carriers. Ear Hear. 2021 Nov-Dec 01;42(6):1525-1543. doi: 10.1097/AUD.0000000000001070. PMID 34369417
- [Derived] JanssensdeVarebeke SPF, Moyaert J, Fransen E, Bulen B, Neesen C, Devroye K, van de Berg R, Pennings RJE, Topsakal V, Vanderveken O, Van Camp G, Van Rompaey V. Genotype-phenotype Correlation Study in a Large Series of Patients Carrying the p.Pro51Ser (p.P51S) Variant in COCH (DFNA9): Part I-A Cross-sectional Study of Hearing Function in 111 Carriers. Ear Hear. 2021 Nov-Dec 01;42(6):1508-1524. doi: 10.1097/AUD.0000000000001099. PMID 34369416